CLINICAL TRIAL: NCT03468257
Title: Testing a Novel Stress-induced Eating Intervention for Cancer Prevention
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never started
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, A. Janet Tomiyama, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 16-000893
Record Dates: First submitted 2018-03-11; First posted 2018-03-16 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: 7-dose Control - Progressive Muscle Relaxation Only; 5-dose - Pairs Progressive Muscle Relaxation With Fruit 5 Consecutive Days; 7-dose - Pairs Progressive Muscle Relaxation With Fruit 7 Consecutive Days; 9-dose - Pairs Progressive Muscle Relaxation With Fruit 9 Consecutive Days

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive Muscle Relaxation only (Active Comparator): Condition 1: 7-dose control - Progressive Muscle Relaxation only
  Interventions: Behavioral: Pavlovian Conditioning
- Pairs Progressive Muscle Relaxation with fruit (Experimental): Condition 2: 5-dose - Pairs Progressive Muscle Relaxation with fruit 5 consecutive days; Condition 3: 7-dose - Pairs Progressive Muscle Relaxation with fruit 7 consecutive days; Condition 4: 9-dose - Pairs Progressive Muscle Relaxation with fruit 9 consecutive days
  Interventions: Behavioral: Pavlovian Conditioning

INTERVENTIONS:
Behavioral: Pavlovian Conditioning — Imagining a stressful event, engaging in progressive muscle relaxation, and eating fruit

SUMMARY:
Subjects will be enrolled in a stress-induced eating intervention with 5, 7, or 9 treatments or control. Treatment will comprise imagining a stressful event, engaging in a stress relief activity (Progressive Muscle Relaxation), and consuming a fruit once per day. There will be one lab visit at baseline in which participants undergo an acute laboratory stressor (i.e., speech and math tasks) and consume food from a buffet. There will be another lab visit at two weeks post-intervention. In the second (and final) lab visit, participants will repeat the acute laboratory stressor (i.e., speech and math tasks) and buffet, and additionally complete questionnaires about their experience in the study.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* fluent in English
* access to an internet-connected device
* reporting a neutral taste and moderate novelty for at least one fruit
* reporting household size-adjusted income less than or equal to 200% of the federal poverty threshold
* perceived stress scale score of 21.82 (1 SD above the national mean)
* BMI 25
* scoring 3.23 on the Dutch Eating Behavior-Emotional Eating Questionnaire

Exclusion Criteria:

* on a diet that would compel them to refrain from eating food in the laboratory buffet
* allergy to any foods presented in the buffet
* selecting a fruit as one or more of top three choices of foods that would make them feel better if stressed

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Healthy Eating Index | 14 days after last dose
  The Healthy Eating Index was developed by the USDA to capture diet quality. The total score is able to capture both the healthiness of fruits and the unhealthiness of classic comfort foods that are high in calories, fat, and sugar.

SECONDARY OUTCOMES:
Calorie intake | 14 days after last dose
  Calorie intake will be recorded across all the foods that the participants choose to eat in the outcome assessment buffet.
Acceptability/Credibility | 14 days after last dose
  The Credibility/Expectancy Questionnaire is a validated measure to access issues of intervention acceptability, credibility, and expectancy.